CLINICAL TRIAL: NCT00021801
Title: Pathways to Tolerance in Human Islet Transplantation
Brief Title: Islet Cell Transplantation Alone and CD34+ Enriched Bone Marrow Cell Infusion in Patients With Diabetes Mellitus: Steroid-Free Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: dk56953 (completed); DK56953-01
Record Dates: First submitted 2001-08-04; First posted 2001-08-06 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type I Diabetes Mellitus; Immunosuppression; Islet Cell Transplant; Percutaneous Transhepatic Portal
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Islets of Langerhans Transplantation

INTERVENTIONS:
Procedure: Islet Cell Transplantation

SUMMARY:
The goal of islet cell transplantation in Type 1 diabetics is to provide those affected with constant normal blood glucose levels, thereby reducing or eliminating altogether the need for injected insulin. This normalization may prevent or slow progression of diabetic complications, result in a healthier lifestyle, and lead to a better quality of life.

Participants who meet the inclusion criteria will undergo an extensive screening process which typically includes a series of blood tests, EKG, chest x-rays, and a psychological evaluation, among others. Those who are eligible for and chose to participate in the trial will receive an islet cell transplant and bone marrow infusion from the same donor, together with following immunosuppressive medications: tacrolimus, sirolimus, daclizumab and infliximab. Because the bone marrow infusion may successfully prevent the transplanted islet cells from rejecting, some participants may be able to stop taking the immunosuppressive medications after a year.

The islet cell transplant is done under local anesthesia in a special procedure radiology room. Several days after the islet cell transplant, the participant is admitted to the hospital as an outpatient in order to receive bone marrow via a simple intra-venous infusion procedure.

All participants will need to be seen at the Diabetes Research Institute after the transplant for follow-up testing and post-islet cell transplant care.

ELIGIBILITY:
Inclusion Criteria:

* Candidates must be between the ages of 18 and 50.
* Candidates must have had insulin-dependent diabetes mellitus (IDDM) for at least 5 years and been under physician care for at least 6 months prior to enrollment in trial.
* Eligible candidates will have poorly controlled IDDM and manifest signs and symptoms severe enough to be incapacitating. These symptoms can include episodes of hypoglycemic unawareness (failure to recognize blood glucose levels < 54 mg/dl) or episodes requiring the assistance of others.
* Candidates may have poor diabetes control despite intensive insulin therapy (HbA1c > 8.0%).
* Creatinine clearance should be > 60 ml/min)
* Body Mass Index should be less than 26
* Women of child-bearing age must have a negative pregnancy test and agree to follow effective contraceptive measures for the duration of the trial.

Exclusion Criteria:

* Previous or concurrent organ transplant
* Previous or concurrent malignancy
* Untreated proliferative diabetic retinopathy
* Unstable cardiovascular status, including positive stress echocardiography (if > age 35)
* Active infections, including x-ray evidence of pulmonary infection
* Peptic ulcer disease, gall stones, or portal hypertension
* Abnormal liver function tests
* Presence of panel reactive antibodies > 20%
* Creatinine clearance < 60 ml/min
* HbA1c > 12%
* Serological evidence of HIV, HbsAg, or HCV
* Anemia (hemoglobin < 12.0)
* Any condition or circumstance, including psychogenic factors, that preclude therapeutic compliance or otherwise make it unsafe to undergo an islet cell transplant.
* PSA > 4 in males

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2000-03; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Alejandro, MD, Principal Investigator — University of Miami Diabetes Research Institute
Locations (1):
- University of Miami Diabetes Research Institute, Miami, Florida, United States

REFERENCES:
- [Background] Alejandro R, Lehmann R, Ricordi C, Kenyon NS, Angelico MC, Burke G, Esquenazi V, Nery J, Betancourt AE, Kong SS, Miller J, Mintz DH. Long-term function (6 years) of islet allografts in type 1 diabetes. Diabetes. 1997 Dec;46(12):1983-9. doi: 10.2337/diab.46.12.1983. PMID 9392484
- [Derived] Tharavanij T, Betancourt A, Messinger S, Cure P, Leitao CB, Baidal DA, Froud T, Ricordi C, Alejandro R. Improved long-term health-related quality of life after islet transplantation. Transplantation. 2008 Nov 15;86(9):1161-7. doi: 10.1097/TP.0b013e31818a7f45. PMID 19005394